CLINICAL TRIAL: NCT05090605
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Breast Cancer in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1186
Record Dates: First submitted 2021-09-25; First posted 2021-10-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: GWAS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with breast cancer
  Interventions: Genetic: DNA analysis
- Control group: Patients without breast cancer
  Interventions: Genetic: DNA analysis

INTERVENTIONS:
Genetic: DNA analysis — GWAS

SUMMARY:
This is a GWAS study that aims to identify possible candidate genes associate to breast cancer by exploring single nucleotide polymorphism (SNP) in a group of breast cancer, in the Kazakh population. The investigators hypothesize that the careful phenotyping of the subject sand matching with increase the power to find SNP significantly associate with breast cancer

DETAILED DESCRIPTION:
A genome-wide association study (GWAS) is an approach used in genetics research to associate specific genetic variations with particular diseases. The method involves scanning the genomes from many different people and looking for genetic markers that can be used to predict the presence of a disease. Once such genetic markers are identified, they can be used to understand how genes contribute to the disease and develop better prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a histologically confirmed diagnosis of breast cancer.
* The age of patients is from 18 to 60 years;
* Persons of Kazakh nationality, whose paternal and maternal grandparents are Kazakhs.
* Persons who are able and willing to provide written informed consent;
* Persons capable and willing to comply with the research protocol;

Exclusion Criteria:

* Persons under 18 and over 60 years old;
* Persons who, in the opinion of the researcher, are mentally or legally incapacitated, which prevents obtaining informed consent;
* Pregnant or lactating women;
* Tuberculosis of any localization in the active phase and in history;
* Severe and decompensated diseases of the liver and kidneys, cardiovascular system;
* Severe and decompensated course of endocrine diseases;
* Lack of histological verification of breast tumor

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: in a group of breast cancer, in the Kazakh population
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with breast cancer | 1 year
  Using GWAS to identify candidate genes associate with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Dilyara Radikovna Kaidarova, M.D, Prof., Academician of the, Study Director — JSC "Kazakh Institute of Oncology and Radiology", Almaty, Kazakhstan; Nazgul Omarbayeva, M.D / PhD, Principal Investigator — JSC "Kazakh Institute of Oncology and Radiology", Almaty, Kazakhstan
Locations (2):
- Kazakhstan (2):
  - JSC "Kazakh Institute of Oncology and Radiology", Almaty
  - JSC "Kazakh Institute of Oncology and Radiology", Almaty, Kazakhstan, Almaty

IPD SHARING:
Plan to Share IPD: Undecided